CLINICAL TRIAL: NCT00790101
Title: An 18-Month, Multicenter, Parallel-Group Study to Determine The Relative Efficacy of Risedronate Versus Raloxifene in Subjects Who Have Discontinued Hormone Replacement Therapy (HRT) for Early Intervention in Osteoporosis
Brief Title: Risedronate vs Raloxifene in Hormone Replacement Therapy Discontinuation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi-Aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HMR4003B_4033
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid; Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): Risedronate 35mg once a week
  Interventions: Drug: Risedronate
- 2 (Active Comparator): Raloxifene 60mg daily
  Interventions: Drug: Raloxifene
- 3 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Risedronate
  Arms: 1
Drug: Raloxifene
  Arms: 2
Other: Placebo
  Arms: 3

SUMMARY:
This is a multi-center, randomized, double-blind, double-dummy study designed to compare the effects of risedronate, raloxifene, and placebo on BMD, bone turnover markers, and other markers of anabolic activity in postmenopausal women who previously received HRT.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal, ambulatory females, "postmenopausal" defined as the absence of menses for at least 12 continuous months)
* In general good health as determined by medical history, physical examination, and laboratory tests
* LS spine BMD T-score between -1.0 and -2.4, inclusive
* At least one analyzable BMD site at both the hip (left or right) and LS spine (at least 3 measurable lumbar spine vertebrae, without fracture or sufficient degenerative disease)
* Currently receiving no medications for the treatment or prevention of osteoporosis
* Had been on continuous HRT for at least 1 year prior to enrollment. The HRT must have ended within 18 months prior to the baseline visit, and the subject must have been off HRT medication for at least 3 months at the time of baseline visit
* Subjects rendered menopausal by surgical procedures between the ages of 55 and 65 years

Exclusion Criteria:

* A history of cancer within 10 years prior to entry into the study, except for relatively "benign" and cured skin cancers such as basal and squamous cell carcinoma
* A history of hyperparathyroidism, hyperthyroidism, osteomalacia, or other metabolic bone disease within one year prior to enrollment
* Any condition or disease that may interfere with the evaluation of at least 3 lumbar vertebrae (not necessarily contiguous), determined in a screening radiograph by a radiologist at the central facility (e.g., confluent aortic calcifications, severe osteoarthritis, spinal fusion, lumbar spine fractures)
* Evidence of clinically significant organic or psychiatric disease on history or physical examination, which in the opinion of the investigator would prevent the patient from completing the study
* Markedly abnormal pretreatment laboratory finds that, in the opinion of the investigator, would prevent the patient from completing the study
* A history of using any of the following medications prior to starting study:
* Any bisphosphonate therapy
* Selective estrogen receptor modulators (SERMs)
* Parathyroid hormone
* Fluorides
* Calcitonin
* Calcitriol (>1.5 mcg/week)
* Corticosteroids on a chronic basis for period equal to or greater then 3 months
* Received a depot injection of >10,000 IU Vitamin D in the past 12 months
* A history of recurrent nephrolithiasis or a history of one episode of nephrolithiasis within 1 year of study entry
* Serum creatinine >1.6 mg/dl
* Unable to sit or stand upright for 30 minutes after taking the morning dose of risedronate
* A history of deep vein thrombosis or other coagulation disorders
* Severe hepatic insufficiency
* A history of hypersensitivity to raloxifene, risedronate, or to drugs with similar chemical structures
* Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult
* Subjects found to have one or more vertebral fractures after completing thoracic and LS spine films
* Subjects who have experienced a low impact fracture related to osteopenia within two years of baseline visit

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Max Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-06; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Compare the effects of risedronate and raloxifene on lumbar spine (LS) bone mineral density (BMD) in osteopenic women previously treated with HRT, who discontinued HRT at least 3 months prior to the study but no greater than 18 mos

SECONDARY OUTCOMES:
Compare the effects of risedronate, raloxifene, and placebo on BMD of the hip

CONTACTS AND LOCATIONS:
Overall Officials: Tara Semanchik, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States